CLINICAL TRIAL: NCT00771641
Title: Phase III Randomized Comparison of Radiotherapy Fractionation in Advanced Squamous Cell Carcinoma of the Head and Neck: Twice-Daily Hyperfractionation vs Split-Course Accelerated Hyperfractionation vs Accelerated Fractionation With Concomitant Boost vs Standard Fractionation
Brief Title: Fractionated Radiation Therapy in Treating Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9003; CDR0000076475
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard Fractionation (Active Comparator): Standard Fractionation: 2 Gy/Fx, Q.D. 5 Days/wk, Total Dose: 70 Gy/35 Fx x 7 wks
  Interventions: Procedure: conventional surgery; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Radiation: radiation therapy
- Hyperfractionation (Experimental): Hyperfractionation: 1.2 Gy/Fx, b.i.d. (> 6 hours apart, 5 days/wk) Total Dose: 81.6 Gy/68 Fx/7 weeks
  Interventions: Procedure: conventional surgery; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Radiation: radiation therapy
- Accelerated Hyperfractionation with split (Experimental): Accelerated Hyperfractionation with split: 1.6 Gy/Fx b.i.d. (> 6 hours apart), 5 days/wk, Total Dose: 67.2 Gy/42 Fx/6 wks with a 2 week rest after 38.4 Gy
  Interventions: Procedure: conventional surgery; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Radiation: radiation therapy
- Accelerated fractionation with concomitant boost (Experimental): Accelerated fractionation with concomitant boost
  Interventions: Procedure: conventional surgery; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy; Radiation: radiation therapy

INTERVENTIONS:
Procedure: conventional surgery
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Patient abstract not available

PURPOSE: Patient abstract not available

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether hyperfractionation and/or accelerated fractionation (split-course or with a concomitant boost) improves the locoregional control rate over standard fractionation radiotherapy in patients with advanced squamous cell carcinomas of the head and neck. II. Determine the disease-free survival and overall survival of these patients treated with different radiotherapy fractionation schemes. III. Determine the acute and late toxicities of each fractionation schedule. IV. Compare the quality of life on the two regimens.

OUTLINE: Randomized study. Arm I: Radiotherapy. Irradiation of primary tumor and involved and at-risk nodal areas using linear accelerators with photon energies of 1.25-6.0 MV (dual energy arrangements may also use a beam greater than 6.0 MV), electrons of 4-25 MV, or Co60. Standard fractionation. Arm II: Radiotherapy. Targets and equipment as in Arm I. Hyperfractionation. Arm III: Radiotherapy. Targets and equipment as in Arm I. Accelerated split-course hyperfractionation. Arm IV: Radiotherapy. Targets and equipment as in Arm I. Accelerated fractionation with concomitant boost.

PROJECTED ACCRUAL: A total of 1,080 patients (270/arm) will be accrued over 5.75 years. If excessive toxicity is noted in any arm after entry of 324 and 634 patients, that arm may be closed.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma of the head and neck, including lymphoepithelioma and anaplastic carcinoma Biopsy from the primary or regional nodes acceptable No adenocarcinomas The following stages and sites are eligible: Stage III/IV oral cavity, including: Anterior 2/3 of the tongue Buccal mucosa Floor of mouth Hard palate Gingiva Retromolar trigone Stage III/IV oropharynx, including: Tonsil and pillars Faucial arch and soft palate Posterolateral pharyngeal walls Stage II/III/IV base of the tongue and hypopharynx Stage III/IV supraglottic larynx, including: Ventricular band Arytenoid Supra- and infrahyoid epiglottis Aryepiglottic fold (tumors at glottic and subglottic sites excluded) Nonpalpable nodes detected only on CT or MRI must be at least 1.0 cm in diameter or contain necrosis to prove N+ disease No metastasis below the clavicle clinically or radiologically

PATIENT CHARACTERISTICS: Age: At least 18 Performance status: Karnofsky 60-100% Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Medically able to withstand radiotherapy No second malignancy within 5 years except nonmelanomatous skin cancer Follow-up by participating radiotherapist required

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to head and neck No planned combined external beam and interstitial boost irradiation Surgery: No prior surgery (other than biopsy) No planned combined pre- or postoperative programs Radical neck dissections allowed if lymph nodes are greater than 3 cm prior to radiotherapy or involvement persists after treatment Resection of persistent disease at the primary site may be performed 6 weeks after completion of radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1113 (Actual)
Dates: Primary Completion 2002-08 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Kian Ang, MD, PhD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- [Background] Gillison ML, Zhang Q, Jordan R, Xiao W, Westra WH, Trotti A, Spencer S, Harris J, Chung CH, Ang KK. Tobacco smoking and increased risk of death and progression for patients with p16-positive and p16-negative oropharyngeal cancer. J Clin Oncol. 2012 Jun 10;30(17):2102-11. doi: 10.1200/JCO.2011.38.4099. Epub 2012 May 7. PMID 22565003
- [Background] Dilling TJ, Bae K, Paulus R, Watkins-Bruner D, Garden AS, Forastiere A, Kian Ang K, Movsas B. Impact of gender, partner status, and race on locoregional failure and overall survival in head and neck cancer patients in three radiation therapy oncology group trials. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):e101-9. doi: 10.1016/j.ijrobp.2011.01.013. Epub 2011 May 5. PMID 21549515
- [Background] Coyne JC, Pajak TF, Harris J, Konski A, Movsas B, Ang K, Watkins Bruner D; Radiation Therapy Oncology Group. Emotional well-being does not predict survival in head and neck cancer patients: a Radiation Therapy Oncology Group study. Cancer. 2007 Dec 1;110(11):2568-75. doi: 10.1002/cncr.23080. PMID 17955501
- [Background] Schumaker L, Nikitakis N, Goloubeva O, Tan M, Taylor R, Cullen KJ. Elevated expression of glutathione S-transferase pi and p53 confers poor prognosis in head and neck cancer patients treated with chemoradiotherapy but not radiotherapy alone. Clin Cancer Res. 2008 Sep 15;14(18):5877-83. doi: 10.1158/1078-0432.CCR-08-0998. PMID 18794100
- [Background] Siddiqui F, Pajak TF, Watkins-Bruner D, Konski AA, Coyne JC, Gwede CK, Garden AS, Spencer SA, Jones C, Movsas B. Pretreatment quality of life predicts for locoregional control in head and neck cancer patients: a radiation therapy oncology group analysis. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):353-60. doi: 10.1016/j.ijrobp.2007.06.024. Epub 2007 Sep 24. PMID 17889449
- [Background] Spiegel D, Kraemer HC. Emotional well-being does not predict survival in head and neck cancer patients: a Radiation Therapy Oncology Group study. Cancer. 2008 May 15;112(10):2326-7; author reply 2327-8. doi: 10.1002/cncr.23435. No abstract available. PMID 18338746
- [Background] Sanabria A, Carvalho AL, Kowalski LP. Is nutrition support related to a poor prognosis in head and neck cancer patients? Thoughts about the secondary analysis of RTOG trial 90-03. Head Neck. 2007 May;29(5):518-9; author reply 519-20. doi: 10.1002/hed.20617. No abstract available. PMID 17390379
- [Background] Konski AA, Pajak T, Movsas B, et al.: Socio-demographic variables influence outcome in Radiation Therapy Oncology Group head and neck trials. [Abstract] Proceedings of the American Society of Clinical Oncology 22 (Suppl 14): A-6043, 529s, 2004.
- [Background] Kumar P, Harris J, Garden AS, et al.: Outcome comparisons of four Radiation Therapy Oncology Group (RTOG) trials in patients with stage IV-T4 head and neck (H/N) cancer: encouraging results using intra-arterial (IA) cisplatin (P) and concurrent radiation therapy (RT). [Abstract] J Clin Oncol 22 (Suppl 14): A-5527, 494s, 2004.
- [Background] Movsas B, Konski A, Pajak T, et al.: Quality of life (QOL) variables influence local regional control in Radiation Therapy Oncology Group (RTOG) headsneck trials (9003 and 9111). [Abstract] Int J Radiat Oncol Biol Phys 60 (1 Suppl 1): A-199, S252, 2004.
- [Background] Owen JB, Grigsby PW, Caldwell TM, Konski AA, Johnson DJ, Demas WF, Movsas B, Jones CU, Wasserman TH. Can costs be measured and predicted by modeling within a cooperative clinical trials group? Economic methodologic pilot studies of the radiation therapy oncology group (RTOG) studies 90-03 and 91-04. Int J Radiat Oncol Biol Phys. 2001 Mar 1;49(3):633-9. doi: 10.1016/s0360-3016(00)00770-7. PMID 11172943
- [Result] Chung CH, Dignam JJ, Hammond ME, Klimowicz AC, Petrillo SK, Magliocco A, Jordan R, Trotti A, Spencer S, Cooper JS, Le QT, Ang KK. Glioma-associated oncogene family zinc finger 1 expression and metastasis in patients with head and neck squamous cell carcinoma treated with radiation therapy (RTOG 9003). J Clin Oncol. 2011 Apr 1;29(10):1326-34. doi: 10.1200/JCO.2010.32.3295. Epub 2011 Feb 28. PMID 21357786
- [Result] Chung CH, Dignam J, Hammond ME, et al.: Association of high Gli1 expression with poor survival in head and neck cancer patients treated with radiation therapy (RTOG 9003). [Abstract] J Clin Oncol 28 (Suppl 15): A-5552, 2010.
- [Result] Konski AA, Winter K, Cole BF, Ang KK, Fu KK. Quality-adjusted survival analysis of Radiation Therapy Oncology Group (RTOG) 90-03: phase III randomized study comparing altered fractionation to standard fractionation radiotherapy for locally advanced head and neck squamous cell carcinoma. Head Neck. 2009 Feb;31(2):207-12. doi: 10.1002/hed.20949. PMID 19107946
- [Result] Le QT, Harris J, Magliocco AM, Kong CS, Diaz R, Shin B, Cao H, Trotti A, Erler JT, Chung CH, Dicker A, Pajak TF, Giaccia AJ, Ang KK. Validation of lysyl oxidase as a prognostic marker for metastasis and survival in head and neck squamous cell carcinoma: Radiation Therapy Oncology Group trial 90-03. J Clin Oncol. 2009 Sep 10;27(26):4281-6. doi: 10.1200/JCO.2008.20.6003. Epub 2009 Aug 10. PMID 19667273
- [Result] Calvin DP, Hammond ME, Pajak TF, Trotti AM, Meredith RF, Rotman M, Jones CU, Byhardt RW, Demas WF, Ang KK, Fu KK; Radiation Therapy Oncology Group 90-03 Trial. Microvessel density >or=60 does not predict for outcome after radiation treatment for locally advanced head and neck squamous cell carcinoma: results of a correlative study from the Radiation Therapy Oncology Group (RTOG) 90-03 Trial. Am J Clin Oncol. 2007 Aug;30(4):406-19. doi: 10.1097/COC.0b013e3180342fd4. PMID 17762442
- [Result] Konski AA, Bhargavan M, Owen J, et al.: Altered fractionated radiotherapy is cost-effective in the treatment of locally advanced head and neck cancer: an economic analysis of Radiation Therapy Oncology Group (RTOG) 90-03. [Abstract] J Clin Oncol 24 (Suppl 18): A-6007, 302s, 2006.
- [Result] Rabinovitch R, Grant B, Berkey BA, Raben D, Ang KK, Fu KK, Cooper JS; Radiation Therapy Oncology Group. Impact of nutrition support on treatment outcome in patients with locally advanced head and neck squamous cell cancer treated with definitive radiotherapy: a secondary analysis of RTOG trial 90-03. Head Neck. 2006 Apr;28(4):287-96. doi: 10.1002/hed.20335. PMID 16287132
- [Result] Pajak TF, Trotti A, Gwede CK, et al.: The TAME risk classification system: acute toxicity burden and IPD analysis of RTOG 90-03. [Abstract] Int J Radiat Oncol Biol Phys 63 (2 Suppl 1): A-217, S131, 2005.
- [Result] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Result] Hammond E, Berkey BA, Fu KK, Trotti A, Meredith RF, Jones CU, Byhardt R, Horwitz EM, Ang KK. P105 as a prognostic indicator in patients irradiated for locally advanced head-and-neck cancer: a clinical/laboratory correlative analysis of RTOG-9003. Int J Radiat Oncol Biol Phys. 2003 Nov 1;57(3):683-92. doi: 10.1016/s0360-3016(03)00642-4. PMID 14529772
- [Result] Konski A, Berkey BA, Kian Ang K, Fu KK. Effect of education level on outcome of patients treated on Radiation Therapy Oncology Group Protocol 90-03. Cancer. 2003 Oct 1;98(7):1497-503. doi: 10.1002/cncr.11661. PMID 14508838
- [Result] Tu X, Berkey BA, Zhang HZ, et al.: Impact of EGFR expression on the response of advanced head and neck carcinomas to concomitant boost radiotherapy in a RTOG phase III trial (90-03). Int J Radiat Oncol Biol Phys 57 (2 Suppl): S157, 2003.
- [Result] Ang KK, Berkey BA, Tu X, Zhang HZ, Katz R, Hammond EH, Fu KK, Milas L. Impact of epidermal growth factor receptor expression on survival and pattern of relapse in patients with advanced head and neck carcinoma. Cancer Res. 2002 Dec 15;62(24):7350-6. PMID 12499279
- [Result] Eldridge B, Rabinovitch R, Berkey BA, et al.: The impact of baseline nutritional support on treatment outcome in patients with locally advanced squamous cell cancer of the head and neck treated with definitive radiotherapy: report of the Radiation Therapy Oncology Group (RTOG) trial 90-03. [Abstract] Int J Radiat Oncol Biol Phys 54(2 suppl 1): A-199, 115, 2002.
- [Result] Konski A, Berkey B, Ang KK, et al.: The effect of education level on outcome of patients treated on Radiation Therapy Oncology Group (RTOG) protocol 90-03. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-992, 2002.
- [Result] Calvin DP, Hammond ME, Pajak TF, et al.: Microvessel density (MVD)> 60 does not predict for outcome in advanced head and neck squamous cell carcinoma (HNSCC): results of a prospective study from the RTOG 90-03 trial. [Abstract] Int J Radiat Oncol Biol Phys 51 (3 suppl 1): A-68, 41, 2001.
- [Result] Fisher J, Scott C, Fu K, et al.: Treatment, patient and tumor characteristics impact quality of life (QOL) in patients with locally advanced head and neck cancer: report of the Radiation Therapy Oncology Group (RTOG) trial 90-03. [Abstract] Int J Radiat Oncol Biol Phys 51 (3 suppl 1): A-174, 98, 2001.
- [Result] Konski AA, Scott CB, Ang KK, et al.: Does dose escalation of radiotherapy (RT) improve quality-adjusted survival (QAS) in unresectable head and neck cancer (HNC) patients (Pts)? Radiation Therapy Oncology Group (RTOG) study 90-03. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-906, 227a, 2001.
- [Result] Konski A, Scott C, Ang KK, et al.: Cost-utility analysis of RTOG 90-03: phase III randomized study comparing altered fractionation to standard fractionation radiotherapy for locally advanced head and neck squamous cell carcinoma. [Abstract] Int J Radiat Oncol Biol Phys 51(3 suppl 1): A-87, 48, 2001.
- [Result] Fisher J, Scott C, Fu K, et al.: Randomized study comparing quality of life between standard fractionation radiotherapy and altered fractionation schemas in patients with locally advanced squamous cell cancer of the head and neck. [Abstract] Proceedings of the International Conference on Head and Neck Cancer A201, 117, 2000.
- [Derived] Mell LK, Shen H, Nguyen-Tan PF, Rosenthal DI, Zakeri K, Vitzthum LK, Frank SJ, Schiff PB, Trotti AM 3rd, Bonner JA, Jones CU, Yom SS, Thorstad WL, Wong SJ, Shenouda G, Ridge JA, Zhang QE, Le QT. Nomogram to Predict the Benefit of Intensive Treatment for Locoregionally Advanced Head and Neck Cancer. Clin Cancer Res. 2019 Dec 1;25(23):7078-7088. doi: 10.1158/1078-0432.CCR-19-1832. Epub 2019 Aug 16. PMID 31420360